CLINICAL TRIAL: NCT07197112
Title: A Clinical Study of the Safety and Efficacy of Gimacabtinib Hydrochloride Tablets in Acute GVHD Patients After Failure of or Intolerance to Ruxolitinib-Based Second-Line Therapy.
Brief Title: Study of Gecacitinib in the Treatment of Acute Graft-Versus-Host Disease After Failure of Ruxolitinib-containing Second-line Therapy
Acronym: GRIT
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RJ-BMT-GvHD-002; Self-funded (Other: Ruijin Hospital)
Record Dates: First submitted 2025-09-19; First posted 2025-09-29 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-08

CONDITIONS: Acute Graft Versus Host Disease Grade II-IV; Acute Graft vs Host Disease
Keywords: gecacitinib; II~IV aGVHD; allogeneic hematopoietic stem cell transplantation; ruxolitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental arm (Experimental): Following enrollment, all subjects are planned to receive gecacitinib for at least 28 days while continuing their existing treatments.
  Interventions: Drug: Gecacitinib

INTERVENTIONS:
Drug: Gecacitinib — Administer 50 mg twice daily for a minimum of 28 days.

SUMMARY:
An open-label, single-arm clinical trial to evaluate the safety and efficacy of gecacitinib tablets in patients with acute graft-versus-host disease (GVHD) who have failed or are intolerant to ruxolitinib-containing second-line therapy.

DETAILED DESCRIPTION:
This is an open-label, single-arm study that plans to enroll 15 subjects with confirmed grade II-IV acute graft-versus-host disease (aGVHD). The primary endpoint is the overall response rate (ORR) on day 28 of gecacitinib treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily signed the informed consent form, with age ≥18 years at the time of ICF signing;
2. Recipients who have undergone non-myeloablative, myeloablative, or reduced-intensity allo-HSCT (allogeneic hematopoietic stem cell transplantation) from any donor source (matched unrelated donor, sibling, or haploidentical) using bone marrow, peripheral blood stem cells, or umbilical cord blood;
3. Complete donor engraftment: donor STR ≥95%, peripheral blood absolute neutrophil count (ANC) >0.5×10⁹/L, platelet count >25×10⁹/L (use of growth factors, transfusion support, etc., is permitted);
4. aGVHD patients who have failed second-line treatment including ruxolitinib, defined as follows:

   * GVHD progression: Progressive GVHD (i.e., an increase in the grading of any organ system or involvement of any new organ) compared to pre-ruxolitinib treatment, after receiving ruxolitinib therapy for ≥5 to 10 days;
   * No response to treatment: Failure to achieve partial response or better improvement in GVHD compared to pre-treatment after at least 14 days of ruxolitinib therapy;
   * Loss of response: Objective worsening of GVHD (manifested as increased grading or new organ involvement) after initial improvement, occurring at any time point;
   * Intolerance: Patients with stable or improving SR-aGVHD who discontinue ruxolitinib due to drug-related toxicity (as assessed by the treating physician).
5. ECOG score: 0-2;
6. Expected survival greater than 4 weeks;
7. Ability to swallow tablets;
8. Ability to comply with study and follow-up procedures.

Exclusion Criteria:

1. Patients who have undergone ≥2 allo-HSCT procedures;
2. Development of SR-aGVHD following unplanned donor lymphocyte infusion (DLI) administered for the treatment of malignant relapse. Note: Patients who received planned DLI as part of the transplant procedure, not intended for managing malignant relapse, may be enrolled;
3. Prior use of ruxolitinib in combination with >1 systemic therapy for steroid-refractory aGVHD;
4. Concurrent use of other JAK inhibitors besides ruxolitinib for treatment. Patients who discontinued JAK inhibitor therapy for aGVHD due to side effects rather than refractoriness are also eligible for the study;
5. Patients with active bleeding;
6. Patients diagnosed with or suspected of having chronic GVHD;
7. Presence of uncontrolled active infection. Uncontrolled active infection is defined as: hemodynamic instability due to sepsis, or worsening of symptoms, signs, or radiographic findings attributable to the infection. Persistent fever without symptoms or with resolving symptoms is not considered an uncontrolled active infection;
8. Patients with unresolved toxicity or complications due to allo-HSCT (excluding aGVHD);
9. Any significant clinical or laboratory abnormality that may affect safety evaluation, such as:

   1. Uncontrolled diabetes (fasting blood glucose >13.9 mmol/L);
   2. Hypertension that cannot be controlled to the following range (systolic blood pressure <160 mmHg, diastolic blood pressure <100 mmHg) with two or more antihypertensive agents;
   3. Peripheral neuropathy (NCI-CTCAE v5.0 Grade 2 or higher).
10. History of New York Heart Association Class III or IV congestive heart failure, uncontrolled or unstable angina, myocardial infarction, cerebrovascular accident, or pulmonary embolism within 6 months prior to screening;
11. Presence of arrhythmia requiring treatment at the time of screening, or patients with QTc interval (QTcB) >480 ms;
12. Impaired renal function at screening (serum creatinine >1.5 × ULN);

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2027-02-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate | Within 28 days of first dose
  Overall Response Rate at Day 28

SECONDARY OUTCOMES:
Non-recurrent Mortality Rate | Week 4, Week 8, Week 12, Week 24
  Non-recurrent Mortality Rate at Week 4, Week 8, Week 12, Week 24

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoxia Hu, MD, Principal Investigator — Ruijin Hospital